CLINICAL TRIAL: NCT01981408
Title: Disposition of [^14C]-LY2801653 Following Oral Administration in Healthy Subjects
Brief Title: A Study of LY2801653 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15283; I3O-EW-JSBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [^14C]-LY2801653 (Experimental): Single oral dose of LY2801653 containing 100 micro curies of radioactivity
  Interventions: Drug: [^14C]-LY2801653

INTERVENTIONS:
Drug: [^14C]-LY2801653 — Administered orally

SUMMARY:
This type of study is called a radiolabeled study. For this study, LY2801653 (study drug) has been specially prepared to contain radiolabeled carbon [^14C]. [^14C] is a naturally occurring radioactive form of the element, carbon. This study will increase understanding about how the drug appears in the blood, urine, and stool after it is administered to healthy people. Information about any side effects that may occur will also be collected. This study will last up to 15 days for each participant, not including screening. Screening is required within 28 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy sterile male and female participants
* Have a body mass index (BMI) of 18.5 to 32.0 kilograms per meter squared (kg/m^2), inclusive

Exclusion Criteria:

* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have consumed herbal supplements, grapefruit juice, grapefruits, grapefruit containing products, Seville orange juice, Seville oranges, star fruit, or star fruit juice within 7 days prior to dosing or intend to consume during the study
* Have donated blood of more than 500 milliliter (mL) within the last month
* Have participated in a [14C]-study within the last 6 months prior to admission for this study
* Exposure to significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)
* Have a defecation pattern less than once per 2 days or acute constipation within 3 weeks of day before dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Urinary and Fecal Excretion of LY2801653 Radioactivity over Time expressed as a Percentage of the Total Radioactive Dose Administered | Pre-dose up to 14 days post dose

SECONDARY OUTCOMES:
Plasma Pharmacokinetics of LY2801653 and Radioactivity Maximum Observed Concentration (Cmax) | Pre-dose up to 14 days post dose
Plasma Pharmacokinetics of LY2801653 and Radioactivity Time of Maximum Concentration (tmax) | Pre-dose up to 14 days post dose
Plasma Pharmacokinetics of LY2801653 and Radioactivity Area Under The Concentration-time Curve from zero to the last timepoint with a measurable Concentration (AUC 0 to tlast) | Pre-dose up to 14 days post dose
Relative Abundance of LY2801653 and the Metabolites of LY2801653 in Urine and Feces | Pre-dose up to 14 days post dose
Relative Abundance of LY2801653 and the Metabolites of LY2801653 in Plasma | Pre-dose up to 14 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States